CLINICAL TRIAL: NCT02751307
Title: Treatment of Metabolic Abnormalities in Patients With Schizophrenia: Adjunctive Low-dose Metformin in Patients With Schizophrenia and Metabolic Abnormalities
Brief Title: Adjunctive Low-dose Metformin in Patients With Schizophrenia and Metabolic Abnormalities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Chun-Hsin Chen, Attending Psychiatrist, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMU-JIRB 201303005
Record Dates: First submitted 2016-04-19; First posted 2016-04-26 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Metabolic Syndrome
Keywords: metformin; clozapine; schizophrenia; metabolic traits
MeSH Terms: conditions — Metabolic Syndrome; Schizophrenia | interventions — Metformin; Clozapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- metformin 500 mg/d; clozapine 100 mg (Active Comparator): In the first week, 500 mg of metformin was administered in the morning. In the second week, the dosage was revised to 500 mg of metformin in the morning and the placebo in the evening. During metformin intervention period, the clozapine dose remained unchanged in these recruited clozapine-treated patients.
  Interventions: Drug: metformin 500 mg; Drug: clozapine 100 mg
- metformin 1000 mg/d; clozapine 100 mg (Active Comparator): In the first week, 500 mg of metformin was administered in the morning. In the second week, 500 mg of metformin twice a day was administered. During metformin intervention period, the clozapine dose remained unchanged in these recruited clozapine-treated patients.
  Interventions: Drug: metformin 500 mg; Drug: clozapine 100 mg
- placebo; clozapine 100 mg (Placebo Comparator): In the first week, one pill of placebo was given and in the second week, placebo BID was given. During metformin intervention period, the clozapine dose remained unchanged in these recruited clozapine-treated patients.
  Interventions: Drug: metformin 500 mg; Drug: clozapine 100 mg

INTERVENTIONS:
Drug: metformin 500 mg — metformin 500 mg QAM for metformin 500 mg/d group; metformin 500 mg 1 BID for metformin 1000 mg/d
  Other Names: Loditon
Drug: clozapine 100 mg — Clozapine dose remained unchanged during metformin intervention period in recruited patients.
  Other Names: Clozaril

SUMMARY:
Metformin has been used for alleviating metabolic abnormalities in patients with schizophrenia. Until now, the lowest dose of metformin to treat metabolic abnormalities in clozapine-treated patients is 1000 mg/d. The aim of this study was to determine whether a lower dosage of metformin, such as 500 mg/d, is effective for improving metabolic profiles in clozapine-treated patients with pre-existing metabolic abnormalities.

Methods:

In this 12-week, randomized, double-blind, placebo-controlled trial, metformin 500 mg/d or 1000 mg/d or a placebo was prescribed to clozapine-treated patients with schizophrenia having pre-existing metabolic abnormalities. The recruited patients underwent physical and laboratory evaluations at week-4, week-8, and week-12.

DETAILED DESCRIPTION:
Methods In this 12-week, randomized, double-blind, placebo-controlled trial, metformin 500 mg/d or 1000 mg/d or placebo was prescribed to clozapine-treated patients with schizophrenia having pre-existing metabolic abnormalities. The study was approved by an institutional review board and was conducted at Taipei Medical University-Wan Fang Hospital and Taipei City Psychiatric Center from May 2013 to January 2015. All clinical investigation had been conducted according to the principles expressed in the Declaration of Helsinki. The investigators screened clozapine-treated patients in the first phase and enrolled eligible patients in this clinical trial. Written informed consent was obtained from all patients before the screening.

Patients in the first-phase screening Patients diagnosed with schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition; aged 20-65 years; and who had taken clozapine for at least 3 months were invited to the first-phase screening. Clinical interviews were conducted, and medical records were evaluated for collecting patient demographics and clinical information, namely diagnosis, age of onset, and dosage of clozapine use.

Measurements The height, BW, waist circumference (WC), and blood pressure (BP) of all patients were measured. The body mass index (BMI) was calculated as the BW in kilograms divided by the square of the height in meters. After overnight fasting, blood was collected for analyzing the fasting plasma glucose (FPG), TG, and high-density lipoprotein cholesterol (HDL-C) levels. Under manufacture's guide, fasting TG, FPG, and HDL-C levels were measured using an automated system (Roche Cobas C501).

Patients in the metformin trial Patients in the first-phase screening were enrolled in the present trial if they had at least one of the following metabolic abnormalities: BMI ≥ 24; WC > 90 cm (men) or 80 cm (women); fasting serum TG level ≥ 150 mg/dL; fasting serum HDL-C level ≤ 40 mg/dL (men) or 50 mg/dL (women); systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg; current use of antihypertensive agents; and FPG level = 100-126 mg/dL. The exclusion criteria were the following: history of diabetes mellitus (DM); current use of hypoglycemic or hypolipidemic agents; pregnancy; allergy to metformin; a creatinine level > 1.4 ng/dL; an abnormal liver function test result; and chronic cardiopulmonary insufficiency.

Trial procedures Patients recruited in the trial were randomized to three groups, metformin 500 mg/d, metformin 1000 mg/d, or placebo. The randomization was conducted by a research assistant, who was blinded to the patient's status. To ensure the concealment of the randomization, the metformin and placebo were provided in coded containers. The appearance of the placebo was identical to that of metformin tablets. All patients, caregivers, and investigators were masked to the randomization.

In the first week, 500 mg of metformin was administered in the morning to the groups of metformin 500 mg/d and 1000 mg/d, and placebo was administered to the placebo group. In the second week, the dosage was revised to 500 mg of metformin in the morning and the placebo in the evening for the group of metformin 500 mg/d, 500 mg of metformin twice a day for the group of metformin 1000 mg/d, and placebo twice daily for the placebo group. For all patients, the clozapine dosage remained unchanged throughout the intervention. The recruited patients underwent physical and laboratory evaluations at week-4, week-8, and week-12.

Statistical analyses The investigators used descriptive statistics for summarizing the baseline clinical characteristics of patients and analysis of variance for examining the differences in these characteristics among all groups. Patients who continued the intervention for at least 4 weeks were included in the analyses. The investigators adopted the last observation carried forward (LOCF) approach for replacing missing data, assuming no change in the missing values of metabolic indices after an event of dropout. Furthermore, for investigating whether repeated measures collected in a longitudinal manner change over time, the investigators first used the paired t test for examining differences between the baseline and follow-up measures. Repeated measure analyses were conducted using 2-way within-subjects analysis of variance for examining group (df = 2, between groups), time (df = 3, within subjects), and interaction (df = 6, interaction between time and groups) effects on the changes in metabolic profiles over time. The analyses were conducted using SPSS Version 20.0 (IBM, Armonk, NY). P < 0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed with schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition
2. aged 20-65 years
3. had taken clozapine for at least 3 months
4. had at least one of the following metabolic abnormalities: BMI ≥ 24; WC > 90 cm (men) or 80 cm (women); fasting serum TG level ≥ 150 mg/dL; fasting serum HDL-C level ≤ 40 mg/dL (men) or 50 mg/dL (women); systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg; current use of antihypertensive agents; and FPG level = 100-126 mg/dL.

Exclusion Criteria:

1. history of diabetes mellitus
2. current use of hypoglycemic or hypolipidemic agents
3. pregnancy
4. allergy to metformin
5. a creatinine level > 1.4 ng/dL
6. an abnormal liver function test result
7. chronic cardiopulmonary insufficiency.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changes in body weight | baseline; week-4; week-8; week-12

SECONDARY OUTCOMES:
Changes in waist circumference | baseline; week-4; week-8; week-12
Changes in blood pressure | baseline; week-4; week-8; week-12
Changes in fasting triglyceride level | baseline; week-4; week-8; week-12
Changes in fasting high-density lipoprotein cholesterol level | baseline; week-4; week-8; week-12
Changes in fasting glucose level | baseline; week-4; week-8; week-12
Changes in scores of positive and negative syndrome scale (PANSS) | baseline; week-4; week-8; week-12
  Recruited patients were interviewed by research assistants to get PANSS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsin Chen, MD, Principal Investigator — Department of Psychiatry, Wan Fang Hospital, Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chiu CC, Lu ML, Huang MC, Chen PY, Lin YK, Lin SK, Chen CH. Effects of Low Dose Metformin on Metabolic Traits in Clozapine-Treated Schizophrenia Patients: An Exploratory Twelve-Week Randomized, Double-Blind, Placebo-Controlled Study. PLoS One. 2016 Dec 14;11(12):e0168347. doi: 10.1371/journal.pone.0168347. eCollection 2016. PMID 27973619